CLINICAL TRIAL: NCT02166047
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Multi-center Study to Evaluate the Safety and Efficacy of GS-9620 for the Treatment of Virally-Suppressed Subjects With Chronic Hepatitis B
Brief Title: Study To Evaluate Safety and Efficacy of Vesatolimod for the Treatment of Chronic Hepatitis B Virus in Virally-Suppressed Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-283-1059; 2014-001400-22 (EudraCT Number); ACTRN12614000628640 (Other: ANZCTR)
Record Dates: First submitted 2014-06-16; First posted 2014-06-18 (Estimated); Results first posted 2020-09-02 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: Chronic Hepatitis B
Keywords: Hepatitis B; HBV; GS-9620; TLR-7 Agonist
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — vesatolimod

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Placebo 4 Weeks (Cohort A) (Placebo Comparator): Placebo tablet once a week for 4 weeks
  Interventions: Drug: Placebo
- Vesatolimod 1 mg 4 Weeks (Cohort A) (Experimental): Vesatolimod 1 mg tablet once a week for 4 weeks
  Interventions: Drug: Vesatolimod
- Vesatolimod 2 mg 4 Weeks (Cohort A) (Experimental): Vesatolimod 2 mg tablet once a week for 4 weeks
  Interventions: Drug: Vesatolimod
- Vesatolimod 4 mg 4 Weeks (Cohort A) (Experimental): Vesatolimod 4 mg tablet once a week for 4 weeks
  Interventions: Drug: Vesatolimod
- Placebo 8 Weeks (Cohort B) (Placebo Comparator): Placebo tablet once a week for 8 weeks
  Interventions: Drug: Placebo
- Vesatolimod 1 mg 8 Weeks (Cohort B) (Experimental): Vesatolimod 1 mg tablet once a week for 8 weeks
  Interventions: Drug: Vesatolimod
- Vesatolimod 2 mg 8 Weeks (Cohort B) (Experimental): Vesatolimod 2 mg tablet once a week for 8 weeks
  Interventions: Drug: Vesatolimod
- Vesatolimod 4 mg 8 Weeks (Cohort B) (Experimental): Vesatolimod 4 mg tablet once a week for 8 weeks
  Interventions: Drug: Vesatolimod
- Placebo 12 Weeks (Cohort C) (Placebo Comparator): Placebo tablet once a week for 12 weeks
  Interventions: Drug: Placebo
- Vesatolimod 1 mg 12 Weeks (Cohort C) (Experimental): Vesatolimod 1 mg tablet once a week for 12 weeks
  Interventions: Drug: Vesatolimod
- Vesatolimod 2 mg 12 Weeks (Cohort C) (Experimental): Vesatolimod 2 mg tablet once a week for 12 weeks
  Interventions: Drug: Vesatolimod
- Vesatolimod 4 mg 12 Weeks (Cohort C) (Experimental): Vesatolimod 4 mg tablet once a week for 12 weeks
  Interventions: Drug: Vesatolimod

INTERVENTIONS:
Drug: Vesatolimod — Vesatolimod tablet administered orally
  Other Names: GS-9620
  Arms: Vesatolimod 1 mg 12 Weeks (Cohort C); Vesatolimod 1 mg 4 Weeks (Cohort A); Vesatolimod 1 mg 8 Weeks (Cohort B); Vesatolimod 2 mg 12 Weeks (Cohort C); Vesatolimod 2 mg 4 Weeks (Cohort A); Vesatolimod 2 mg 8 Weeks (Cohort B); Vesatolimod 4 mg 12 Weeks (Cohort C); Vesatolimod 4 mg 4 Weeks (Cohort A); Vesatolimod 4 mg 8 Weeks (Cohort B)
Drug: Placebo — Placebo to match vesatolimod tablet administered orally
  Arms: Placebo 12 Weeks (Cohort C); Placebo 4 Weeks (Cohort A); Placebo 8 Weeks (Cohort B)

SUMMARY:
The primary objectives of this study are to evaluate the safety, tolerability, and efficacy of vesatolimod in participants with chronic hepatitis B (CHB) infection currently being treated with oral antivirals (OAV).

Participants will be randomized in 3 sequential cohorts (Cohorts A, B, and C). Within each cohort, participants will be randomized in a 1:3:3:3 ratio to placebo or one of the doses of vesatolimod (1, 2, or 4 mg).

ELIGIBILITY:
Key Inclusion Criteria:

* Must have the ability to understand and sign a written informed consent form; consent must be obtained prior to initiation of study procedures
* Documented evidence of CHB infection (eg, hepatitis B surface antigen [HBsAg] positive for more than 6 months) with detectable HBsAg levels at screening
* Have been on approved HBV OAV treatment for ≥ 1 year prior to screening, with HBV DNA below lower limit of quantitation (LLOQ), measured at least once, 6 or more months prior to screening, and HBV DNA < 20 IU/mL at screening
* Currently taking an approved HBV OAV (tenofovir, entecavir, adefovir, lamivudine, or telbivudine, either as single agents or in combination) with no change in regimen for 3 months prior to screening
* Willing to provide blood sample for toll-like receptor 7 (TLR-7) and interleukin 28 B (IL28B) single-nucleotide polymorphism (SNP) assessment
* Must be willing and able to comply with all study requirements

Key Exclusion Criteria:

* Extensive bridging fibrosis or cirrhosis
* Laboratory parameters not within defined thresholds for neutropenia, anemia, thrombocytopenia, leukopenia, or other evidence of inadequate liver function
* Coinfection with hepatitis C virus (HCV), HIV, or hepatitis D virus (HDV)
* Evidence of hepatocellular carcinoma
* Malignancy within 5 years prior to screening, with the exception of specific cancers that are cured by surgical resection (basal cell skin cancer, etc.). Participants under evaluation for possible malignancy are not eligible.
* Significant cardiovascular, pulmonary, or neurological disease
* Any of the following conditions that may worsen in response to interferon (IFN):

  * Autoimmune disease (eg, lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, sarcoidosis, moderate or severe psoriasis)
  * Poorly controlled diabetes mellitus
  * Significant psychiatric disorders
  * Thyroid disorder (unless controlled under treatment)
  * Significant pulmonary diseases (eg, chronic obstructive pulmonary disease)
  * Retinal disease
  * Immunodeficiency disorders
* Received solid organ or bone marrow transplant
* Received prolonged therapy with immunomodulators (eg, corticosteroids) or biologics (eg, monoclonal Ab, interferon) within 3 months of screening
* Use of another investigational agents within 3 months of screening
* Current alcohol or substance abuse judged by the investigator to potentially interfere with compliance
* Females who are pregnant or may wish to become pregnant during the study

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2014-06-30 (Actual); Primary Completion 2016-05-11 (Actual); Study Completion 2016-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (18):
- United States (8):
  - Los Angeles, California
  - San Diego, California
  - San Francisco, California
  - San Jose, California
  - Honolulu, Hawaii
  - Boston, Massachusetts
  - Detroit, Michigan
  - Flushing, New York
- Canada (3):
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Toronto, Ontario
- Italy (4):
  - San Giovanni Rotondo, FG
  - Milan
  - Parma
  - Pisa
- Rotterdam, Netherlands
- Auckland, New Zealand
- Seoul, South Korea

REFERENCES:
- [Result] Boni C, Vecchi A, Rossi M, Laccabue D, Giuberti T, Alfieri A, Lampertico P, Grossi G, Facchetti F, Brunetto MR, Coco B, Cavallone D, Mangia A, Santoro R, Piazzolla V, Lau A, Gaggar A, Subramanian GM, Ferrari C. TLR7 Agonist Increases Responses of Hepatitis B Virus-Specific T Cells and Natural Killer Cells in Patients With Chronic Hepatitis B Treated With Nucleos(T)Ide Analogues. Gastroenterology. 2018 May;154(6):1764-1777.e7. doi: 10.1053/j.gastro.2018.01.030. Epub 2018 Jan 31. PMID 29378197
- [Result] Janssen HLA, Brunetto MR, Kim YJ, Ferrari C, Massetto B, Nguyen AH, Joshi A, Woo J, Lau AH, Gaggar A, Subramanian GM, Yoshida EM, Ahn SH, Tsai NCS, Fung S, Gane EJ. Safety, efficacy and pharmacodynamics of vesatolimod (GS-9620) in virally suppressed patients with chronic hepatitis B. J Hepatol. 2018 Mar;68(3):431-440. doi: 10.1016/j.jhep.2017.10.027. Epub 2017 Dec 11. PMID 29104121

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States, Canada, Italy, South Korea, The Netherlands, and New Zealand. The first participant was screened on 30 June 2014. The last study visit occurred on 20 October 2016.
Pre-assignment Details: All participants continued their approved HBV oral antiviral therapy (tenofovir disoproxil fumarate (TDF), entecavir (ETV), adefovir, lamivudine, or telbivudine, either as single agents or in combination) throughout the study.
  200 participants were screened.
Period: Overall Study
Arm/Group | Vesatolimod 1 mg 4 Weeks (Cohort A) | Vesatolimod 2 mg 4 Weeks (Cohort A) | Vesatolimod 4 mg 4 Weeks (Cohort A) | Placebo 4 Weeks (Cohort A) | Vesatolimod 1 mg 8 Weeks (Cohort B) | Vesatolimod 2 mg 8 Weeks (Cohort B) | Vesatolimod 4 mg 8 Weeks (Cohort B) | Placebo 8 Weeks (Cohort B) | Vesatolimod 1 mg 12 Weeks (Cohort C) | Vesatolimod 2 mg 12 Weeks (Cohort C) | Vesatolimod 4 mg 12 Weeks (Cohort C) | Placebo 12 Weeks (Cohort C)
Started | 16 | 15 | 16 | 5 | 18 | 17 | 17 | 5 | 16 | 17 | 14 | 6
Completed | 16 | 14 | 14 | 5 | 17 | 17 | 15 | 5 | 16 | 17 | 12 | 6
Not Completed | 0 | 1 | 2 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Participant | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vesatolimod 1 mg 4 Weeks (Cohort A) | Vesatolimod 2 mg 4 Weeks (Cohort A) | Vesatolimod 4 mg 4 Weeks (Cohort A) | Placebo 4 Weeks (Cohort A) | Vesatolimod 1 mg 8 Weeks (Cohort B) | Vesatolimod 2 mg 8 Weeks (Cohort B) | Vesatolimod 4 mg 8 Weeks (Cohort B) | Placebo 8 Weeks (Cohort B) | Vesatolimod 1 mg 12 Weeks (Cohort C) | Vesatolimod 2 mg 12 Weeks (Cohort C) | Vesatolimod 4 mg 12 Weeks (Cohort C) | Placebo 12 Weeks (Cohort C) | Total
Number analyzed (Participants) | 16 | 15 | 16 | 5 | 18 | 17 | 17 | 5 | 16 | 17 | 14 | 6 | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (7.3) | 50 (11.2) | 47 (10.0) | 53 (5.3) | 51 (8.2) | 44 (9.0) | 44 (11.1) | 53 (5.4) | 48 (9.8) | 48 (9.7) | 50 (11.6) | 46 (10.9) | 48 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 4 | 1 | 9 | 4 | 4 | 1 | 5 | 2 | 3 | 0 | 39
  Male | 15 | 10 | 12 | 4 | 9 | 13 | 13 | 4 | 11 | 15 | 11 | 6 | 123
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 13 | 10 | 12 | 4 | 15 | 15 | 16 | 4 | 9 | 8 | 9 | 2 | 117
  Race: Native Hawaiian or Pacific Islander | 1 | 2 | 3 | 0 | 2 | 1 | 1 | 0 | 7 | 8 | 5 | 4 | 34
  Race: White | 2 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 7
  Race: Black or African American | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Race: Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Not Hispanic or Latino | 16 | 15 | 16 | 5 | 18 | 17 | 17 | 5 | 16 | 17 | 14 | 6 | 162
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 8 | 3 | 3 | 0 | 4 | 5 | 2 | 0 | 2 | 2 | 2 | 2 | 33
  Italy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 9 | 2 | 28
  Netherlands | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 6
  New Zealand | 4 | 2 | 6 | 3 | 1 | 3 | 0 | 0 | 3 | 2 | 0 | 0 | 24
  South Korea | 0 | 0 | 0 | 0 | 7 | 4 | 9 | 3 | 1 | 2 | 1 | 1 | 28
  United States | 4 | 10 | 7 | 2 | 3 | 4 | 5 | 1 | 1 | 3 | 2 | 1 | 43
Serum Hepatitis B Surface Antigen (HBsAg) Level [Mean (Standard Deviation); unit: log10 IU/mL] | 2.8 (0.88) | 3.1 (0.59) | 3.0 (0.70) | 3.1 (0.69) | 3.1 (0.62) | 3.0 (0.69) | 3.1 (0.90) | 2.7 (0.73) | 3.3 (0.45) | 3.0 (0.54) | 3.0 (0.69) | 2.4 (1.01) | 3.0 (0.70)
Serum HBsAg Level Categories [Count of Participants; unit: Participants]
  ≤ 5000 IU/mL | 13 | 13 | 13 | 4 | 15 | 15 | 14 | 5 | 14 | 15 | 13 | 5 | 139
  > 5000 IU/mL | 3 | 2 | 3 | 1 | 3 | 2 | 3 | 0 | 2 | 2 | 1 | 1 | 23
Hepatitis B Envelope Antigen (HBeAg) Status [Count of Participants; unit: Participants]
  Negative | 12 | 11 | 12 | 4 | 13 | 14 | 14 | 5 | 13 | 14 | 12 | 4 | 128
  Positive | 4 | 4 | 4 | 1 | 5 | 3 | 3 | 0 | 3 | 3 | 2 | 2 | 34

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Serum Hepatitis B Surface Antigen (HBsAg) Level at Week 24
Description: A mixed effect model for repeated measures (MMRM) was used to analyze HBsAg change from baseline, which included treatment, baseline HBsAg level (> 5000 IU/mL or ≤ 5000 IU/mL), HBeAg baseline status (positive or negative), visit and treatment-by-visit interaction as fixed effect and visit as repeated measurement.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set (participants who were randomized and received at least 1 dose of study drug) with available data were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: log10 IU/mL
Arm/Group | Vesatolimod 1 mg 4 Weeks (Cohort A) | Vesatolimod 2 mg 4 Weeks (Cohort A) | Vesatolimod 4 mg 4 Weeks (Cohort A) | Placebo 4 Weeks (Cohort A) | Vesatolimod 1 mg 8 Weeks (Cohort B) | Vesatolimod 2 mg 8 Weeks (Cohort B) | Vesatolimod 4 mg 8 Weeks (Cohort B) | Placebo 8 Weeks (Cohort B) | Vesatolimod 1 mg 12 Weeks (Cohort C) | Vesatolimod 2 mg 12 Weeks (Cohort C) | Vesatolimod 4 mg 12 Weeks (Cohort C) | Placebo 12 Weeks (Cohort C)
Number analyzed (Participants) | 16 | 14 | 15 | 5 | 17 | 17 | 16 | 5 | 16 | 17 | 12 | 6
log10 IU/mL | -0.011 [-0.054 to 0.031] | 0.033 [-0.012 to 0.079] | -0.018 [-0.062 to 0.026] | -0.035 [-0.109 to 0.040] | -0.081 [-0.145 to -0.016] | -0.081 [-0.147 to -0.014] | -0.082 [-0.148 to -0.015] | -0.163 [-0.281 to -0.045] | -0.015 [-0.057 to 0.027] | 0.000 [-0.041 to 0.042] | 0.000 [-0.046 to 0.047] | 0.001 [-0.057 to 0.058]
Statistical Analysis 1: Comparison: Vesatolimod 1 mg 4 Weeks (Cohort A) vs Placebo 4 Weeks (Cohort A); Test type: Superiority; p = 0.590, MMRM — P-value between vesatolimod and placebo was not adjusted for multiplicity due to exploratory nature of the study; Least Squares (LS) Mean Difference = 0.023, 95% CI 2-sided [-0.061 to 0.108]
Statistical Analysis 2: Comparison: Vesatolimod 2 mg 4 Weeks (Cohort A) vs Placebo 4 Weeks (Cohort A); Test type: Superiority; p = 0.120, MMRM — P-value between vesatolimod and placebo was not adjusted for multiplicity due to exploratory nature of the study; LS Mean Difference = 0.068, 95% CI 2-sided [-0.018 to 0.154]
Statistical Analysis 3: Comparison: Vesatolimod 4 mg 4 Weeks (Cohort A) vs Placebo 4 Weeks (Cohort A); Test type: Superiority; p = 0.701, MMRM — P-value between vesatolimod and placebo was not adjusted for multiplicity due to exploratory nature of the study; LS Mean Difference = 0.017, 95% CI 2-sided [-0.069 to 0.102]
Statistical Analysis 4: Comparison: Vesatolimod 1 mg 8 Weeks (Cohort B) vs Placebo 8 Weeks (Cohort B); Test type: Superiority; p = 0.210, MMRM — P-value between vesatolimod and placebo was not adjusted for multiplicity due to exploratory nature of the study; LS Mean Difference = 0.082, 95% CI 2-sided [-0.046 to 0.210]
Statistical Analysis 5: Comparison: Vesatolimod 2 mg 8 Weeks (Cohort B) vs Placebo 8 Weeks (Cohort B); Test type: Superiority; p = 0.207, MMRM — P-value between vesatolimod and placebo was not adjusted for multiplicity due to exploratory nature of the study; LS Mean Difference = 0.082, 95% CI 2-sided [-0.046 to 0.210]
Statistical Analysis 6: Comparison: Vesatolimod 4 mg 8 Weeks (Cohort B) vs Placebo 8 Weeks (Cohort B); Test type: Superiority; p = 0.216, MMRM — P-value between vesatolimod and placebo was not adjusted for multiplicity due to exploratory nature of the study; LS Mean Difference = 0.081, 95% CI 2-sided [-0.048 to 0.210]
Statistical Analysis 7: Comparison: Vesatolimod 1 mg 12 Weeks (Cohort C) vs Placebo 12 Weeks (Cohort C); Test type: Superiority; p = 0.652, MMRM — P-value between vesatolimod and placebo was not adjusted for multiplicity due to exploratory nature of the study; LS Mean Difference = -0.015, 95% CI 2-sided [-0.081 to 0.051]
Statistical Analysis 8: Comparison: Vesatolimod 2 mg 12 Weeks (Cohort C) vs Placebo 12 Weeks (Cohort C); Test type: Superiority; p = 0.994, MMRM — P-value between vesatolimod and placebo was not adjusted for multiplicity due to exploratory nature of the study; LS Mean Difference = -0.000, 95% CI 2-sided [-0.066 to 0.065]
Statistical Analysis 9: Comparison: Vesatolimod 4 mg 12 Weeks (Cohort C) vs Placebo 12 Weeks (Cohort C); Test type: Superiority; p = 0.996, MMRM — P-value between vesatolimod and placebo was not adjusted for multiplicity due to exploratory nature of the study; LS Mean Difference = -0.000, 95% CI 2-sided [-0.069 to 0.069]

2. Secondary Outcome: Composite Endpoint Measuring the Percentage of Participants With Hepatitis B Envelope Antigen (HBeAg) Loss and Seroconversion at Week 24
Description: HBeAg loss was defined as qualitative HBeAg result changing from positive at baseline to negative at any postbaseline visit within the targeted time window.
  HBeAg seroconversion was defined as qualitative hepatitis B envelope antibody (HBeAb) result changing from negative at baseline to positive at any postbaseline visit within the targeted time window.
  Participants who had missing information were assumed to have no HBeAg loss and no HBeAg seroconversion.
Time Frame: Week 24
Population: Participants in the Full Analysis Set with HBeAg+ at Baseline were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Vesatolimod 1 mg 4 Weeks (Cohort A) | Vesatolimod 2 mg 4 Weeks (Cohort A) | Vesatolimod 4 mg 4 Weeks (Cohort A) | Placebo 4 Weeks (Cohort A) | Vesatolimod 1 mg 8 Weeks (Cohort B) | Vesatolimod 2 mg 8 Weeks (Cohort B) | Vesatolimod 4 mg 8 Weeks (Cohort B) | Placebo 8 Weeks (Cohort B) | Vesatolimod 1 mg 12 Weeks (Cohort C) | Vesatolimod 2 mg 12 Weeks (Cohort C) | Vesatolimod 4 mg 12 Weeks (Cohort C) | Placebo 12 Weeks (Cohort C)
Number analyzed (Participants) | 4 | 4 | 4 | 1 | 5 | 3 | 3 | 0 | 3 | 3 | 2 | 2
percentage of participants | 0.0 | 0.0 | 0.0 | 0.0 | 20.0 | 0.0 | 0.0 |  | 0.0 | 0.0 | 0.0 | 0.0

3. Secondary Outcome: Composite Endpoint Measuring the Percentage of Participants With Hepatitis B Envelope Antigen (HBeAg) Loss and Seroconversion at Week 48
Description: HBeAg loss was defined as qualitative HBeAg result changing from positive at baseline to negative at any postbaseline visit within the targeted time window.
  HBeAg seroconversion was defined as qualitative hepatitis B envelope antibody (HBeAb) result changing from negative at baseline to positive at any postbaseline visit within the targeted time window.
  Participants who had missing information were assumed to have no HBeAg loss and no HBeAg seroconversion.
  Only participants who were HBeAg+ at baseline were included.
Time Frame: Week 48
Population: Participants in the Full Analysis Set with HBeAg+ at Baseline were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Vesatolimod 1 mg 4 Weeks (Cohort A) | Vesatolimod 2 mg 4 Weeks (Cohort A) | Vesatolimod 4 mg 4 Weeks (Cohort A) | Placebo 4 Weeks (Cohort A) | Vesatolimod 1 mg 8 Weeks (Cohort B) | Vesatolimod 2 mg 8 Weeks (Cohort B) | Vesatolimod 4 mg 8 Weeks (Cohort B) | Placebo 8 Weeks (Cohort B) | Vesatolimod 1 mg 12 Weeks (Cohort C) | Vesatolimod 2 mg 12 Weeks (Cohort C) | Vesatolimod 4 mg 12 Weeks (Cohort C) | Placebo 12 Weeks (Cohort C)
Number analyzed (Participants) | 4 | 4 | 4 | 1 | 5 | 3 | 3 | 0 | 3 | 3 | 2 | 2
percentage of participants | 0.0 | 0.0 | 0.0 | 0.0 | 20.0 | 0.0 | 0.0 |  | 33.3 | 0.0 | 0.0 | 0.0

4. Secondary Outcome: Composite Endpoint Measuring the Percentage of Participants With HBsAg Loss and Seroconversion at Week 24
Description: HBsAg loss was defined as qualitative HBsAg result changing from positive at baseline to negative at any postbaseline visit within the targeted time window.
  HBsAg seroconversion was defined as qualitative hepatitis B surface antibody (HBsAb) result changing from negative at baseline to positive at any postbaseline visit within the targeted time window.
  Participants who had missing information were assumed to have no HBsAg loss and no HBsAg seroconversion.
Time Frame: Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Vesatolimod 1 mg 4 Weeks (Cohort A) | Vesatolimod 2 mg 4 Weeks (Cohort A) | Vesatolimod 4 mg 4 Weeks (Cohort A) | Placebo 4 Weeks (Cohort A) | Vesatolimod 1 mg 8 Weeks (Cohort B) | Vesatolimod 2 mg 8 Weeks (Cohort B) | Vesatolimod 4 mg 8 Weeks (Cohort B) | Placebo 8 Weeks (Cohort B) | Vesatolimod 1 mg 12 Weeks (Cohort C) | Vesatolimod 2 mg 12 Weeks (Cohort C) | Vesatolimod 4 mg 12 Weeks (Cohort C) | Placebo 12 Weeks (Cohort C)
Number analyzed (Participants) | 16 | 15 | 16 | 5 | 18 | 17 | 17 | 5 | 16 | 17 | 14 | 6
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Composite Endpoint Measuring the Percentage of Participants With HBsAg Loss and Seroconversion at Week 48
Description: as for outcome 4
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Vesatolimod 1 mg 4 Weeks (Cohort A) | Vesatolimod 2 mg 4 Weeks (Cohort A) | Vesatolimod 4 mg 4 Weeks (Cohort A) | Placebo 4 Weeks (Cohort A) | Vesatolimod 1 mg 8 Weeks (Cohort B) | Vesatolimod 2 mg 8 Weeks (Cohort B) | Vesatolimod 4 mg 8 Weeks (Cohort B) | Placebo 8 Weeks (Cohort B) | Vesatolimod 1 mg 12 Weeks (Cohort C) | Vesatolimod 2 mg 12 Weeks (Cohort C) | Vesatolimod 4 mg 12 Weeks (Cohort C) | Placebo 12 Weeks (Cohort C)
Number analyzed (Participants) | 16 | 15 | 16 | 5 | 18 | 17 | 17 | 5 | 16 | 17 | 14 | 6
percentage of participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

6. Secondary Outcome: Change From Baseline in Serum HBsAg Level at Week 4
Time Frame: Baseline; Week 4
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Vesatolimod 1 mg 4 Weeks (Cohort A) | Vesatolimod 2 mg 4 Weeks (Cohort A) | Vesatolimod 4 mg 4 Weeks (Cohort A) | Placebo 4 Weeks (Cohort A) | Vesatolimod 1 mg 8 Weeks (Cohort B) | Vesatolimod 2 mg 8 Weeks (Cohort B) | Vesatolimod 4 mg 8 Weeks (Cohort B) | Placebo 8 Weeks (Cohort B) | Vesatolimod 1 mg 12 Weeks (Cohort C) | Vesatolimod 2 mg 12 Weeks (Cohort C) | Vesatolimod 4 mg 12 Weeks (Cohort C) | Placebo 12 Weeks (Cohort C)
Number analyzed (Participants) | 15 | 14 | 14 | 5 | 18 | 17 | 17 | 5 | 16 | 17 | 13 | 6
log10 IU/mL | -0.009 (0.0505) | 0.025 (0.0514) | -0.008 (0.0516) | -0.017 (0.0600) | -0.003 (0.0574) | 0.014 (0.0794) | -0.001 (0.0436) | 0.046 (0.0648) | -0.034 (0.0375) | -0.023 (0.0529) | -0.001 (0.0627) | -0.041 (0.0955)

7. Secondary Outcome: Change From Baseline in Serum HBsAg Level at Week 8
Time Frame: Baseline; Week 8
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Vesatolimod 1 mg 4 Weeks (Cohort A) | Vesatolimod 2 mg 4 Weeks (Cohort A) | Vesatolimod 4 mg 4 Weeks (Cohort A) | Placebo 4 Weeks (Cohort A) | Vesatolimod 1 mg 8 Weeks (Cohort B) | Vesatolimod 2 mg 8 Weeks (Cohort B) | Vesatolimod 4 mg 8 Weeks (Cohort B) | Placebo 8 Weeks (Cohort B) | Vesatolimod 1 mg 12 Weeks (Cohort C) | Vesatolimod 2 mg 12 Weeks (Cohort C) | Vesatolimod 4 mg 12 Weeks (Cohort C) | Placebo 12 Weeks (Cohort C)
Number analyzed (Participants) | 16 | 13 | 15 | 4 | 17 | 17 | 17 | 4 | 16 | 17 | 12 | 6
log10 IU/mL | -0.029 (0.0666) | 0.002 (0.0544) | -0.035 (0.0649) | -0.013 (0.0440) | 0.000 (0.0442) | 0.006 (0.0772) | 0.020 (0.0596) | 0.006 (0.0600) | -0.021 (0.0376) | -0.033 (0.0487) | -0.013 (0.0426) | -0.019 (0.0483)

8. Secondary Outcome: Change From Baseline in Serum HBsAg Level at Week 12
Time Frame: Baseline; Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Vesatolimod 1 mg 4 Weeks (Cohort A) | Vesatolimod 2 mg 4 Weeks (Cohort A) | Vesatolimod 4 mg 4 Weeks (Cohort A) | Placebo 4 Weeks (Cohort A) | Vesatolimod 1 mg 8 Weeks (Cohort B) | Vesatolimod 2 mg 8 Weeks (Cohort B) | Vesatolimod 4 mg 8 Weeks (Cohort B) | Placebo 8 Weeks (Cohort B) | Vesatolimod 1 mg 12 Weeks (Cohort C) | Vesatolimod 2 mg 12 Weeks (Cohort C) | Vesatolimod 4 mg 12 Weeks (Cohort C) | Placebo 12 Weeks (Cohort C)
Number analyzed (Participants) | 14 | 14 | 15 | 5 | 17 | 17 | 16 | 5 | 16 | 16 | 12 | 6
log10 IU/mL | -0.050 (0.0755) | 0.017 (0.0646) | -0.004 (0.0546) | -0.023 (0.0623) | -0.031 (0.0817) | -0.005 (0.0843) | -0.021 (0.0716) | -0.020 (0.0666) | -0.023 (0.0545) | -0.034 (0.0549) | -0.010 (0.0621) | -0.024 (0.0661)

9. Secondary Outcome: Change From Baseline in Serum HBsAg Level at Week 48
Time Frame: Baseline; Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Vesatolimod 1 mg 4 Weeks (Cohort A) | Vesatolimod 2 mg 4 Weeks (Cohort A) | Vesatolimod 4 mg 4 Weeks (Cohort A) | Placebo 4 Weeks (Cohort A) | Vesatolimod 1 mg 8 Weeks (Cohort B) | Vesatolimod 2 mg 8 Weeks (Cohort B) | Vesatolimod 4 mg 8 Weeks (Cohort B) | Placebo 8 Weeks (Cohort B) | Vesatolimod 1 mg 12 Weeks (Cohort C) | Vesatolimod 2 mg 12 Weeks (Cohort C) | Vesatolimod 4 mg 12 Weeks (Cohort C) | Placebo 12 Weeks (Cohort C)
Number analyzed (Participants) | 16 | 13 | 14 | 4 | 17 | 16 | 15 | 5 | 16 | 17 | 12 | 6
log10 IU/mL | -0.048 (0.1054) | -0.055 (0.1400) | -0.071 (0.0857) | -0.067 (0.0831) | -0.035 (0.0923) | -0.024 (0.0679) | -0.114 (0.2169) | -0.324 (0.6811) | -0.083 (0.0858) | -0.071 (0.1076) | -0.054 (0.0715) | -0.063 (0.1011)

ADVERSE EVENTS:
Time Frame: Adverse Events: First dose date up to Week 12 plus 30 days; All-Cause Mortality: Baseline up to Week 48
Description: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Arm/Group | Vesatolimod 1 mg 4 Weeks (Cohort A) | Vesatolimod 2 mg 4 Weeks (Cohort A) | Vesatolimod 4 mg 4 Weeks (Cohort A) | Placebo 4 Weeks (Cohort A) | Vesatolimod 1 mg 8 Weeks (Cohort B) | Vesatolimod 2 mg 8 Weeks (Cohort B) | Vesatolimod 4 mg 8 Weeks (Cohort B) | Placebo 8 Weeks (Cohort B) | Vesatolimod 1 mg 12 Weeks (Cohort C) | Vesatolimod 2 mg 12 Weeks (Cohort C) | Vesatolimod 4 mg 12 Weeks (Cohort C) | Placebo 12 Weeks (Cohort C)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15 | 0/16 | 0/5 | 0/18 | 0/17 | 0/17 | 0/5 | 0/16 | 0/17 | 0/14 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/16 | 1/15 | 1/16 | 0/5 | 0/18 | 0/17 | 0/17 | 0/5 | 0/16 | 1/17 | 1/14 | 0/6
Other Adverse Events (participants affected / at risk) | 10/16 | 12/15 | 13/16 | 4/5 | 12/18 | 7/17 | 10/17 | 4/5 | 12/16 | 12/17 | 9/14 | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vesatolimod 1 mg 4 Weeks (Cohort A) (N=16) | Vesatolimod 2 mg 4 Weeks (Cohort A) (N=15) | Vesatolimod 4 mg 4 Weeks (Cohort A) (N=16) | Placebo 4 Weeks (Cohort A) (N=5) | Vesatolimod 1 mg 8 Weeks (Cohort B) (N=18) | Vesatolimod 2 mg 8 Weeks (Cohort B) (N=17) | Vesatolimod 4 mg 8 Weeks (Cohort B) (N=17) | Placebo 8 Weeks (Cohort B) (N=5) | Vesatolimod 1 mg 12 Weeks (Cohort C) (N=16) | Vesatolimod 2 mg 12 Weeks (Cohort C) (N=17) | Vesatolimod 4 mg 12 Weeks (Cohort C) (N=14) | Placebo 12 Weeks (Cohort C) (N=6)
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vesatolimod 1 mg 4 Weeks (Cohort A) (N=16) | Vesatolimod 2 mg 4 Weeks (Cohort A) (N=15) | Vesatolimod 4 mg 4 Weeks (Cohort A) (N=16) | Placebo 4 Weeks (Cohort A) (N=5) | Vesatolimod 1 mg 8 Weeks (Cohort B) (N=18) | Vesatolimod 2 mg 8 Weeks (Cohort B) (N=17) | Vesatolimod 4 mg 8 Weeks (Cohort B) (N=17) | Placebo 8 Weeks (Cohort B) (N=5) | Vesatolimod 1 mg 12 Weeks (Cohort C) (N=16) | Vesatolimod 2 mg 12 Weeks (Cohort C) (N=17) | Vesatolimod 4 mg 12 Weeks (Cohort C) (N=14) | Placebo 12 Weeks (Cohort C) (N=6)
Ear swelling (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mouth cyst (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 5 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 4 | 3 | 3 | 1 | 2 | 0 | 2 | 1 | 4 | 2 | 1 | 1
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Feeling hot (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 4 | 0 | 3 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal dryness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 0 | 3 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 3 | 1
Thirst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vessel puncture site bruise (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Oral pustule (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Root canal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Blood pressure abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 1 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 3 | 2 | 2 | 6 | 2 | 4 | 2 | 4 | 3 | 3 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Initial insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Middle insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Micturition frequency decreased (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nail growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years